CLINICAL TRIAL: NCT04929431
Title: Validation of an Algorithm to Predict the Ventilatory Threshold for Exercise Intensity Prescription in Patients With Cardiovascular Disease
Brief Title: Validation of an Algorithm to Predict the Ventilatory Threshold
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: University of Brasilia (Other); University of Bern (Other); Universitaire Ziekenhuizen KU Leuven (Other); University of Siena (Other); Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Prof. Dr., Hasselt University
Other Study IDs: VT algorithm validation
Record Dates: First submitted 2021-05-18; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the current study was to develop an algorithm which has the ability to accurately predict the first and second ventilatory threshold and in cardiovascular disease patients and to guide in proper exercise intensity determination. This would then help, at least in part, to overcome the lack of access to metabolic carts or cardiopulmonary exercise test, and/or methodological difficulties with ventilatory threshold determination in these patients.

DETAILED DESCRIPTION:
Design

This study is composed out of two sub studies: 1. Generation/creation of VT prediction algorithm, and 2. Validation of this algorithm in independent laboratories.

Sub study 1: Generation/creation of VT prediction algorithm

From April 2015 up to July 2020, data from CVD (risk) patients (e.g. obesity, diabetes, coronary artery disease or heart failure) were collected from in light of research studies. All participants signed an informed consent explaining the nature and risks of CPET, and allowing us to use anonymized data for the analyses of their CPET at entry of cardiovascular rehabilitation or an exercise intervention. These data have been published in previous publications.

Sub study 2: Validation of the algorithm in independent laboratories

From April 2015 up to July 2020, data from CVD (risk) patients (e.g. obesity, diabetes, coronary artery disease or heart failure) were collected in light of research studies. All participants signed an informed consent (approved by the ethics committees of the local hospitals or research laboratories) explaining the nature and risks of CPET, and allowing us to use anonymized data for the analyses of their CPET at entry of CR or an exercise intervention. These data have been published in previous publications

ELIGIBILITY:
Inclusion Criteria:

* CVD patients (eg obesity, diabetes, coronary heart disease, heart failure)

Exclusion Criteria:

* No present CVD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From April 2015 up to July 2020, data from CVD (risk) patients (e.g. obesity, diabetes, coronary artery disease or heart failure) were collected from Jessa hospital, Hasselt, Belgium, and Hasselt university, Faculty of Rehabilitation Sciences, Hasselt, Belgium, in light of research studies. All participants signed an informed consent (approved by the ethical committees of Jessa hospital Hasselt and/or Hasselt University) explaining the nature and risks of CPET, and allowing us to use anonymized data for the analyses of their CPET at entry of CR or an exercise intervention
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Duration during cardiopulmonary exercise testing | Baseline - day 1
  Test duration (min)
Workload during cardiopulmonary exercise testing | Baseline - day 1
  Peak workload (watt)
Heart rate during cardiopulmonary exercise testing | Baseline - day 1
  Peak heart rate (bpm)
Oxygen uptake during cardiopulmonary exercise testing | Baseline - day 1
  Maximal oxygen uptake (ml/kg/min)
Heart rate in rest during cardiopulmonary exercise testing | Baseline - day 1
  Resting heart rate (bpm)

SECONDARY OUTCOMES:
Hypertension (in mmHg) | Baseline
  Blood pressure measurement with a automatic blood pressure cuff.
Dyslipdemia (in mg/dl) | Baseline
  Blood lipid concentration in mg/dl
Diabetes (mg/dl) | Baseline
  Glucose concentration in the blood in mg/dl
Obesity | Baseline
  Presence of obesity determined by the BMI (see below)
Smoking | Baseline
  Presence of smoking by questionnaire (yes/no)
Medication intake | Baseline
  Information regarding medication intake will be retrospectively extracted by personal communication with the subject
Cardiovascular surgery | Baseline
  Information regarding cardiovascular surgery will be extracted by personal communication with the subject
Age in years | Baseline
  Age in years will be retrospectively extracted from the databank
Gender (m/f) | Baseline
  Gender in m/f will be retrospectively extracted from the databank
Length in meters | Baseline
  Length in meter will be retrospectively extracted from the databank
Weight in kg | Baseline
  Weight in kg will be retrospectively extracted from the databank
BMI (kg/m^2) | Baseline
  Weight (in kg) and height (in m) will be combined to assess BMI (in kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, Prof.dr, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided